CLINICAL TRIAL: NCT01622933
Title: A Phase I Trial Testing Multiple Antigen-Engineered DC Followed by IFNa2b Boost for Immunization of HLA-Unrestricted Melanoma Patients
Brief Title: Multiple Antigen-Engineered DC Vaccine for Melanoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Lisa H. Butterfield, Ph.D. (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, Lisa H. Butterfield, Ph.D., Professor of Medicine, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 09-021; 1P50CA121973-01A1 (NIH)
Record Dates: First submitted 2012-06-14; First posted 2012-06-19 (Estimated); Last update posted 2017-08-31 (Actual); Status verified 2016-05

CONDITIONS: Melanoma
Keywords: melanoma; recurrent; metastatic
MeSH Terms: conditions — Melanoma; Recurrence; Neoplasm Metastasis | interventions — Introns

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vaccine + IFN (Experimental): Subjects will receive the investigational vaccine, intradermally, every other week for a total of 3 vaccines. Approximately 30 days after the last vaccine subjects will receive IFN intravenously 5 days a week for 4 weeks.
  Leukapheresis will be required to be performed for each subject to be able to produce the investigational vaccine and for research testing. Leukapheresis and biopsies will be performed before the first vaccine, after the 3rd vaccine, and after the IFN treatment.
  Interventions: Biological: DC Vaccine + IFN
- Vaccine only (Experimental): Subjects will receive the investigational vaccine, intradermally, every other week for a total of 3 vaccines.
  Leukapheresis will be required to be performed for each subject to be able to produce the investigational vaccine and for research testing. Leukapheresis and biopsies will be performed before the first vaccine, after the 3rd vaccine, and again approximately 2 months after the last vaccine.
  Interventions: Biological: AdVTMM2/DC Vaccination

INTERVENTIONS:
Biological: DC Vaccine + IFN — Vaccine: The dose target is 1x10e7 AdVTMM2/DC per intradermal injection, or lower dose per sponsor's discretion.
  IFN: 20 MU/m²/d (rounded to the nearest 1.0 million unit) administered IV x 5 consecutive days out of 7 (M-F) every week x 4 weeks.
  Other Names: Interferon Alfa - 2b; Intron A; IFN-alpha 2b; NSC #377523; IFNα; AdVTMM2/DC Vaccination
  Arms: Vaccine + IFN
Biological: AdVTMM2/DC Vaccination — Vaccine: The dose target is 1x10e7 AdVTMM2/DC per intradermal injection.If cell counts are below the target, as few as 5x10e6 AdVTMM2/DC may be administered. However, at the discretion of the sponsor and/or the treating physician, a lower dose of DC that fulfills all of the other criteria for release may be administered on a case by case basis. If this occurs a dose exception form will be completed by the IMCPL, signed by the treating physician and filed in the subjects research records.
  Arms: Vaccine only

SUMMARY:
This clinical trial is to determine if the addition of a standard of care drug, interferon-alfa 2b (IFN), with an investigation vaccine will have any affect on the immune system and/or your cancer. The investigational vaccine will be made with genes that are specific to melanoma and will be given intradermally (i.d.) every two weeks for a total of 3 vaccines.

After the vaccines, subjects will be randomized to either receive a boost of high dose IFN or no boost. IFN will be administered intravenously (into a vein) for 5 consecutive days (Monday through Friday) every week for 4 weeks. Administration will begin approximately 30 days (± 7 days) after the 3rd vaccine. The first dose of IFNα2b may begin within 10 business days of randomization. All subsequent procedure dates for Group A will be based on the date of the first dose of IFNα2b.

DETAILED DESCRIPTION:
This is a Phase I, single site study to evaluate the immunological effects of autologous DC transduced with the MART-1, tyrosinase and MAGE-A6 (melanoma associated antigens, MAA) genes in 30 subjects with recurrent, unresectable stage III, IV metastatic melanoma (M1a, M1b, M1c). AdVTMM2-transduced DC, 10e7, will be given intradermally (i.d.) every two weeks for a total of 3 vaccines.

After the DC vaccines, subjects will be randomized to either receive a boost of high dose IFNa2b or no boost.

Subjects randomized to receive the IFNa2b boost will receive Interferon-a2b, 20 MU/m2/d (rounded to the nearest 1 million units) administered intravenously for 5 consecutive days (Monday through Friday) every week for 4 weeks (induction). Administration will begin approximately 30 days (± 7 days) after the 3rd vaccine. The first dose of IFNα2b may begin within 10 business days of randomization. All subsequent procedure dates for Group A will be based on the date of the first dose of IFNα2b..

The end-points of this study are local and systemic toxicity, immunological response, generation of determinant spreading and anti-tumor immunity, and clinical response.

ELIGIBILITY:
Inclusion Criteria:

* Ability and willing to give consent
* Patients age 18 and older with recurrent, inoperable stage III, IV, M1a, b or c melanoma (any tumor thickness and any number of lymph node involvement, and in-transit metastases, or distant metastases) (AJCC).

Previously treated with any form of therapy (including chemotherapy, radiation therapy, immunotherapy or surgery) for either metastatic, relapsed, or primary melanoma are eligible for this trial, provided the previous treatment was completed > 30 days prior to enrollment.

* Patients should have at least 2 subcutaneous, intracutaneous, and accessible tumor deposits, lymph node or other site available for biopsy purposes.
* Both men and women may be enrolled. Premenopausal females must have a negative pregnancy test prior to treatment and lactating females will have to discontinue breast feeding to be eligible.
* ECOG Performance Status of 0 or 1.
* No previous evidence of class 3 or greater New York Heart Association cardiac insufficiency or coronary artery disease.
* No previous evidence of opportunistic infection.
* Adequate baseline hematological and organ function as assessed by the following laboratory values within 28 days prior to study entry:

Hemoglobin >/=9 g/dL Granulocytes >/=2,000/mm3 Lymphocytes >/=1000/mm3 Platelets >100,000/mm3 Serum Creatinine </=1.5 X the ULN AST, ALT, GGT, CPK, LDH, Alk phos </=2.5 X the ULN Serum Bilirubin </=1.5 X ULN In addition to study entry, the above hematological and organ function lab values along with the ECOG PS must be met prior to starting IFNα treatment.

* Subjects must have normal coagulation parameters as measured by PT/PTT,unless the subject is on an anticoagulation therapy.

Exclusion Criteria:

* Females of child-bearing potential (pre-menopausal) must have a negative serum beta-HCG pregnancy test at screening.
* Subjects with acute infection: any acute viral, bacterial, or fungal infection which requires specific therapy. Acute therapy must have been completed more than 14 days prior to study treatment.
* Hep B & C and HIV-infected patients, due to concerns in the ability to stimulate an effective immune response (determined by historical medical data).
* Subjects with acute medical problems such as ischemic heart or lung disease that may be considered an unacceptable anesthetic or operative risk.
* Subjects with any underlying conditions which would contraindicate therapy with study treatment (or allergies to reagents).
* Subjects with organ allografts.
* Subjects must be free of known brain metastases by contrast-enhanced CT/MRI scans or have successfully-treated brain metastases and be asymptomatic for more than 1 month.
* Patients requiring immunosuppressive therapy for comorbid conditions.
* Concomitant Medication and Treatment: All allowed medications or treatments should be kept to a minimum and recorded. All questions regarding concomitant medications should be referred to the Investigator.
* Long term concurrent medications and/or treatments Not Allowed: Corticosteroids, chemotherapy, cyclosporin A. Short term (approximately 1 week) use of topical, low-dose or inhaled steroids may be allowed at the discretion of the investigator. Injectables not allowed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2012-06; Primary Completion 2016-05 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Safety | 2 years
  Types of adverse events associated with this Multiple Antigen-Engineered DC vaccine at the injection site and systemically.

SECONDARY OUTCOMES:
Immunological response (antigen-specific T cell activation) | 2 years
  Antigen-specific T cell activation will be monitored.

CONTACTS AND LOCATIONS:
Overall Officials: John M Kirkwood, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh Cancer Institute, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Derived] Butterfield LH, Vujanovic L, Santos PM, Maurer DM, Gambotto A, Lohr J, Li C, Waldman J, Chandran U, Lin Y, Lin H, Tawbi HA, Tarhini AA, Kirkwood JM. Multiple antigen-engineered DC vaccines with or without IFNalpha to promote antitumor immunity in melanoma. J Immunother Cancer. 2019 Apr 24;7(1):113. doi: 10.1186/s40425-019-0552-x. PMID 31014399